CLINICAL TRIAL: NCT00397566
Title: Randomized, Placebo-Controlled, Ascending Multiple Dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of BMS-707035 in HIV-1 Infected Subjects
Brief Title: A Multiple Ascending Dose Study of BMS-707035 in HIV-1 Infected Subjects
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AI441-008
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: HIV Infections
Keywords: HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Integrase Inhibitors; BMS-707035

INTERVENTIONS:
Drug: HIV Integrase Inhibitor (BMS-707035)

SUMMARY:
The purpose of this clinical research study is to assess the safety, pharmacokinetics and pharmacodynamics of BMS-707035 in subjects infected with HIV-1

ELIGIBILITY:
Inclusion Criteria:

* HIV-1-infected subjects with CD4+ lymphocyte count ≥ 200 cells/mm3 and with plasma HIV-1 RNA ≥ 5000 copies/mL who have not been on antiretroviral (ARV) therapy for ≥ 8 weeks or who are naive to ARV, and who are otherwise medically stable as determined by medical history, physical examination, 12 lead electrocardiogram, and clinical laboratory evaluations will be eligible to participate in the study. In addition, subjects must have had no prior exposure to the Integrase Inhibitor class of compounds.
* Female subjects must not be nursing, pregnant, or of childbearing potential

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To assess the antiviral activity of selected doses of BMS-707035 administered orally to HIV-1 infected subjects for 10 days.

SECONDARY OUTCOMES:
Safety and tolerability with 10 days of dosing
Effect on QTc intervals
Effect on CD4+, CD8+, and CD8+CD38+ lymphocyte
Pharmacokinetics of multiple doses of BMS-707035 in HIV-1 infected subjects
Assess relationship of EC90 and exposures of BMS-707035 to the magnitude of change in viral loads
Assess plasma protein binding and intracellular concentration in PBMC for BMS-707035